CLINICAL TRIAL: NCT05449574
Title: Sensory Integration Disorders in Multiple Sclerosis
Brief Title: Sensory Integration Disorders in Patients With MS Including Disease Advancement and Relapses in the Last Year
Status: Completed | Type: Observational
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Sponsor
Other Study IDs: PUM
Record Dates: First submitted 2022-06-29; First posted 2022-07-08 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-06

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis;; Sensory integration; relapses; the advancement of the disease
MeSH Terms: conditions — Multiple Sclerosis; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- people with MS: People with MS with relapsing-remitting form
  Interventions: Diagnostic Test: Scale for the Assessment of Sensory Integration in Adults
- healthy people: people from the age of 30-45 years old
  Interventions: Diagnostic Test: Scale for the Assessment of Sensory Integration in Adults

INTERVENTIONS:
Diagnostic Test: Scale for the Assessment of Sensory Integration in Adults — In people with MS and people with health of similar age, a test was performed to assess sensory integration in adults

SUMMARY:
the aim of the study was to assess the occurrence of sensory integration disorders in people with SI depending on the stage of the disease and relapses in the last year;analysis of sensory integration disorders in patients with Ms and healthy people

DETAILED DESCRIPTION:
141 patients diagnosed with RRSM were enrolled in the study. The control group consisted of 72 healthy people. The Sensory Integration Assessment Scale in Adults (SPD) was used to test sensory integration, and an original questionnaire was carried out containing information on age, gender, frequency of relapses in the last year, and duration of the disease.

ELIGIBILITY:
Inclusion Criteria:

* health of a person
* aged 30-45 years
* without diagnosed disorders of sensory integration and MS

Exclusion Criteria:

* diagnosed disorders of sensory integration
* diagnosed with Ms

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients diagnosed with relapsing-remitting MS were qualified for the study; aged 30 to 45
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-06-27 (Actual)

PRIMARY OUTCOMES:
sensory integration disorders and relapses in the last year | 1 year
  Patients with MS were divided into two groups, with relapses in the last year and without relapses. In each group, ters were performed to assess sensory integration in adults. To study SI disorders, the Daniel Travis questionnaire was used to study SI disorders in people over 18 years of age based on the guidelines of the American Society of SI Disorders in Adults. The following domains were distinguished: general sensory processing (OP, 9 items), sensory hypersensitivity (NS, 26 items), hypersensitivity / sensory exploration (PS, 20 items), sensory discrimination (DS, 26 items), motor skills (ZM, 19 items ) and socio-emotional disorders (SE, 22 items). Each symptom was assessed by the participant on a 5-point Likert scale from 0 (never occurred) to 4 (repeats regularly). If the problem occurred in the past, the respondent entered the letter P. The sum obtained by adding values in each of the domains indicated the severity of SI disorders in a given domain.
Sensory integration disorders and the degree of disease severity | 1 Day
  MS patients were divided into two groups with EDSS up to 2.5 points and below. In both groups, sensory integration disorders were checked using a scale to assess sensoryintegration in adults. To study SI disorders, the Daniel Travis questionnaire was used to study SI disorders in people over 18 years of age based on the guidelines of the American Society of SI Disorders in Adults. The following domains were distinguished: general sensory processing (OP, 9 items), sensory hypersensitivity (NS, 26 items), hypersensitivity / sensory exploration (PS, 20 items), sensory discrimination (DS, 26 items), motor skills (ZM, 19 items ) and socio-emotional disorders (SE, 22 items). Each symptom was assessed by the participant on a 5-point Likert scale from 0 (never occurred) to 4 (repeats regularly). If the problem occurred in the past, the respondent entered the letter P. The sum obtained by adding values in each of the domains indicated the severity of SI disorders in a given domain.
Comparing the test group with the control group | 1 Day
  The results of the scale tests were compared to the sensory integration test in the test group and the control group. To study SI disorders, the Daniel Travis questionnaire was used to study SI disorders in people over 18 years of age based on the guidelines of the American Society of SI Disorders in Adults. The following domains were distinguished: general sensory processing (OP, 9 items), sensory hypersensitivity (NS, 26 items), hypersensitivity / sensory exploration (PS, 20 items), sensory discrimination (DS, 26 items), motor skills (ZM, 19 items ) and socio-emotional disorders (SE, 22 items). Each symptom was assessed by the participant on a 5-point Likert scale from 0 (never occurred) to 4 (repeats regularly). If the problem occurred in the past, the respondent entered the letter P. The sum obtained by adding values in each of the domains indicated the severity of SI disorders in a given domain.

CONTACTS AND LOCATIONS:
Overall Officials: Wioletta Pawlukowska, dr hab., Study Chair — Department of Neurology, Pomeranian Medical University, Szczecin, Poland
Locations (1):
- Departmen of Neurology, Szczecin, Unii Lubelskiej, Poland

IPD SHARING:
Plan to Share IPD: No